CLINICAL TRIAL: NCT06383741
Title: Forecast of Functional Outcome and Impact of Anti Factor Xa-levels in Patients With Intracerebral Haemorrhage Related to Direct Factor Xa Inhibitors - a Multi-center Cohort Study
Brief Title: Predicting Outcomes in ICH Patients on Direct Factor Xa Inhibitors
Acronym: FIRE-Xa
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00541
Record Dates: First submitted 2024-01-08; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Intra Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICH study cohort: Patients with intracerebral haemorrhage associated with factor Xa-inhibitor treatment treated at one of the participating centres.

SUMMARY:
This study focuses on direct factor Xa inhibitors (apixaban, edoxaban, rivaroxaban) and the thrombin inhibitor dabigatran, commonly used for stroke prevention in atrial fibrillation. Despite lower intracranial bleeding risks with these drugs, around 0.2-1.0% of patients annually experience intracranial hemorrhage (ICH), predominantly intracerebral.

Treatment options for factor-Xa inhibitor-associated ICH, such as prothrombin complex concentrate (PCC) and andexanet alfa, lack direct comparison evidence except for ongoing trials like ANNEXA-I. This trial assesses hemostatic efficacy and 30-day functional outcomes but leaves gaps regarding anticoagulant activity's role and long-term effects, especially in patients presenting late after drug intake.

The measurement of anti-FXa levels helps guide decisions, yet their link to hematoma expansion remains unknown. Efforts to streamline measurement within 30 minutes for acute decisions have shown variability in levels, with some patients exhibiting high levels even beyond 12 hours post-intake. This lack of data poses challenges, particularly for patients potentially benefiting from treatment beyond the current strict time window.

Early hematoma expansion strongly predicts poor outcomes, but preventing it faces challenges like recurrent events (up to 5% by 3 months) and rehabilitation intensity, potentially negating its benefits. The ANNEXA-I trial evaluates short-term outcomes, highlighting the need for additional data to comprehend long-term ICH prognosis.

The study's objectives involve linking hematoma expansion to anti-FXa levels, determining late-presenting patients' risk of expansion, and identifying predictors of favorable outcomes at 3, 6, and 12 months. Primary endpoints include functional outcomes, while secondary ones encompass expansion rates, anticoagulant activity, and various events at 12 months.

This research aims to bridge gaps in understanding factor-Xa inhibitor-related ICH, addressing both immediate and prolonged outcomes to enhance clinical decision-making.

DETAILED DESCRIPTION:
The utilization of direct oral anticoagulants (DOACs), such as factor Xa inhibitors (apixaban, edoxaban, rivaroxaban) and the thrombin inhibitor dabigatran, has emerged as a pivotal strategy for preventing stroke in patients with atrial fibrillation and thromboembolic diseases. While the risk of intracranial bleeding is notably lower (by about 50%) with DOACs in comparison to Vitamin K antagonists, a fraction of patients (0.2-1.0% annually) still experiences intracranial hemorrhages, primarily intracerebral. Notably, based on data from the Swiss Stroke Registry spanning 2014 to 2019, 9.1% of patients admitted to stroke units or centers for intracerebral hemorrhage (ICH) had prior DOAC therapy. This incidence continues to rise, with 95% of DOAC-associated intracerebral hemorrhages occurring during factor Xa inhibitor therapy.

Treatment strategies for factor Xa inhibitor-associated intracerebral hemorrhage encompass prothrombin complex concentrate (PCC) and the specific reversal agent andexanet alfa. However, the available evidence relies on observational cohort studies and independent patient samples, lacking direct comparative trials. The ongoing randomized controlled trial, ANNEXA-I, aims to assess the efficacy of andexanet alfa compared to standard care. The primary outcome includes hemostatic efficacy measured by imaging within a 12-hour window and functional outcomes evaluated at 30 days. While ANNEXA-I anticipates providing valuable insights into factor Xa-associated intracerebral hemorrhage treatment, significant aspects concerning the role of anticoagulant activity, particularly in patients presenting late after their last dosage intake, and long-term outcomes will remain unanswered.

Assessing anticoagulant activity through anti-FXa levels remains integral yet inconclusive regarding its correlation with hematoma expansion risk. Despite streamlined anti-FXa level measurements at the investigators' institution, heterogeneity in these levels persists, including elevated levels (>100ng/ml) observed even beyond 12 hours post-intake. Notably, the inclusion criteria for ANNEXA-I predominantly consider the time since the last intake (≤15 hours) of factor Xa inhibitors, often omitting anti-FXa level measurements. This oversight might exclude a subgroup of patients who could potentially benefit from andexanet alfa treatment beyond the current strict time window.

Early hematoma expansion significantly impacts outcomes; however, challenges such as recurrent events and rehabilitation intensity may dilute the benefits of preventing hematoma expansion. ANNEXA-I primarily focuses on short-term outcomes, necessitating additional data to comprehend long-term prognoses post intracerebral hemorrhage.

This research aims to establish associations between hematoma expansion and anti-FXa levels, identify risks in late-presenting patients, and predict favorable outcomes at 3, 6, and 12 months. Primary endpoints include functional outcomes, while secondary endpoints involve expansion rates, anticoagulant activity, and various events at the 12-month mark. The comprehensive analysis seeks to bridge gaps in understanding intracerebral hemorrhages associated with DOACs, guiding clinical decisions for both immediate and extended prognoses.

ELIGIBILITY:
Inclusion Criteria:

* Imaging proven intracerebral haemorrhage
* Prior therapy with a factor Xa-inhibitor (apixaban, edoxaban or rivaroxaban), not paused for medical/non-medical reasons for more than 48 hours prior to symptom onset
* Drug-specific calibrated anti-FXa levels measured on admission
* Informed consent (by patient, next-of-kin or deferred consent)

Exclusion Criteria:

* Additional treatment with Vitamin K antagonist or dabigatran

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals admitted to stroke units or stroke centers who experienced intracranial bleeding while on prior direct oral anticoagulant (DOAC) therapy, specifically factor Xa inhibitors such as apixaban, edoxaban, rivaroxaban, and the direct thrombin inhibitor dabigatran. These patients suffered from direct factor Xa inhibitor-associated intracerebral haemorrhage (ICH).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Good functional outcome | At 3 months
  Good functional outcome: defined as mRS 0-3
Good functional outcome | At 6 months
  Good functional outcome: defined as mRS 0-3
Good functional outcome | At 12 months
  Good functional outcome: defined as mRS 0-3

SECONDARY OUTCOMES:
Haematoma expansion | Up to 72hours after baseline imaging
  Haematoma expansion: defined as +33% or 6ml increase between baseline and follow-up imaging
Number of patients with significant anticoagulant activity arriving late | At baseline visit (i.e. hospitalisation)
  Number of patients with significant anticoagulant activity arriving late: defined as last drug intake >12 hours/unknown at hospital arrival and anti-FXa-levels >75ng/ml
Absolute haematoma expansion (in ml) between baseline and follow-up imaging | At 3 and 12 months follow-up hospital visit
  Absolute haematoma expansion (in ml) between baseline and follow-up imaging
Symptomatic haematoma expansion | At 3 and 12 months follow-up hospital visit
  Defined as any increase in volume and decrease in neurological function of >4 points on the NIHSS; investigators are asked whether there is a causal relation between haematoma expansion and functional deterioration
Resumption of anticoagulant therapy after haemorrhage | At 3, 6 and 12 months
  Percentage of patients resuming anticoagulant therapy after haemorrhage
Patients living at home | At 3, 6 and 12 months
  Percentage of patients with the capacity to independently live at home
Functionally independent patients (mRS 0-2) | At 3, 6 and 12 months
  Frequency of functional independence based on mRS after ICH
Excellent outcome (mRS 0-1) | At 3, 6 and 12 months
  Frequency of excellent outcome based on mRS after ICH
Arterial and venous events at 12 months | At 12 months
  Recorded events of arterial and venous complications

CONTACTS AND LOCATIONS:
Overall Officials: David J. Seiffge, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Insel Gruppe AG, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided